CLINICAL TRIAL: NCT00061542
Title: Safety and Efficacy Study of BETOPTIC S 0.25% and Timolol Gel-forming Solution 0.25% and 0.5% in Pediatric Patients With Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-01-01
Record Dates: First submitted 2003-05-28; First posted 2003-05-30 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2008-08

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Betaxolol

ARMS (3):
- Betaxolol (Experimental): Two doses daily for 12 weeks
  Interventions: Drug: BETOPTIC S (betaxolol HCl)
- TGFS 0.25% (Experimental): Two doses daily for 12 weeks
  Interventions: Drug: Timolol Gel-forming Solution (TGFS)
- TGFS 0.5% (Experimental): Two doses daily for 12 weeks
  Interventions: Drug: Timolol Gel-forming Solution (TGFS)

INTERVENTIONS:
Drug: BETOPTIC S (betaxolol HCl) — betaxolol HC)
  Arms: Betaxolol
Drug: Timolol Gel-forming Solution (TGFS) — timolol maleate 0.25% and 0.5%
  Arms: TGFS 0.25%; TGFS 0.5%

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of BETOPTIC S and Timolol Gel-forming solution in pediatric patients. Patients will dose with study drug at 8 am and 8 pm daily for twelve weeks. Patients will have vision tested, slit lamp exam, blood pressure and pulse checks at each visit. Patients will have a dilated fundus exam and corneal measurements taken at first and last visit.

ELIGIBILITY:
INCLUSION:

* Children 5 years old and younger
* require treatment for glaucoma or ocular hypertension
* whose vision is 20/80 or better
* have a cup-to-disc ratio of 0.8 or less

EXCLUSION:

* do not have abnormal fixation
* IOP greater than 36 mm Hg
* significant retinal disease
* penetrating keratoplasty
* severe ocular pathology
* optic atrophy
* eye surgery in the past 30 days
* cardiovascular abnormalities
* hypersensitivity to beta blockers

Ages: 1 Week to 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2003-01; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in IOP | Up to Week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Call Center, Fort Worth, Texas, United States

REFERENCES:
- [Result] Plager DA, Whitson JT, Netland PA, Vijaya L, Sathyan P, Sood D, Krishnadas SR, Robin AL, Gross RD, Scheib SA, Scott H, Dickerson JE; BETOPTIC S Pediatric Study Group. Betaxolol hydrochloride ophthalmic suspension 0.25% and timolol gel-forming solution 0.25% and 0.5% in pediatric glaucoma: a randomized clinical trial. J AAPOS. 2009 Aug;13(4):384-90. doi: 10.1016/j.jaapos.2009.04.017. PMID 19683191